CLINICAL TRIAL: NCT03579654
Title: A Phase 2, Randomized Study of Proscavax, a PSA/IL-2/GM-CSF Vaccine, in Treatment-naive Patients With Clinically Localized Prostate Cancer Versus an Active Surveillance Strategy
Brief Title: Study of Proscavax Vaccine in Patients With Localized Prostate Cancer vs Active Surveillance
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: OncBioMune Pharmaceuticals (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: O17-11110
Record Dates: First submitted 2018-06-06; First posted 2018-07-06 (Actual); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Prostate Cancer
Keywords: Prostate Specific Antigen; Immunotherapy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 - Proscavax vaccine treatment (Experimental): In this arm, during the first 4 months of induction treatment, 6 doses of the Proscavax vaccine will be administered intradermally at weeks 1, 2, 3, 7, 11, and 15, followed by maintenance booster injections once every month which will alternate between low dose IL-2 alone (at weeks 19, 27 and 35) and Proscavax vaccine (at weeks 23, 31, 39) for 6 months.
  Interventions: Biological: Proscavax
- Arm 2 - Active Surveillance (No Intervention): In this arm, patients will undergo active surveillance and will not receive any Proscavax vaccine treatment.

INTERVENTIONS:
Biological: Proscavax — Proscavax is a prostate cancer vaccine which combines the prostate antigen PSA with immune stimulatory cytokines (IL-2 and GM-CSF).
  Arms: Arm 1 - Proscavax vaccine treatment

SUMMARY:
This study will evaluate the safety and efficacy of a prostate cancer vaccine named Proscavax (Prostate-specific antigen(PSA) / Interleukin-2(IL-2) / Granulocyte-macrophage colony-stimulating factor(GM-CSF)) in patients with localized prostate cancer. The goal of the study is to determine if vaccine administration results in a change in the rate of prostate cancer progression when compared to a no-treatment control group of active surveillance patients.

The researchers are interested in evaluating the proportion of participants with prostate cancer progression at 2 years following administration of Proscavax or active surveillance, the effect of the vaccine on prostate-specific antigen (PSA) doubling time and the assessment of adverse events in these patients.

Eligible patients in this study will include men who are 18 years and older and who have a previously untreated early stage prostate cancer regardless of the date of diagnosis.

DETAILED DESCRIPTION:
This study will have 2 arms and patients will be randomized 2:1 into the Proscavax treatment arm (Arm 1) versus the active surveillance arm (Arm 2).

In study Arm 1, 6 doses of the vaccine will be administered intradermally at weeks 1, 2, 3, 7, 11, and 15, followed by maintenance booster injections once every month which will alternate between low dose IL-2 alone (at weeks 19, 27 and 35) and Proscavax vaccine (at weeks 23, 31, 39) for 6 months.

In study Arm 2, patients will undergo active surveillance and will not receive any Proscavax vaccine treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed adenocarcinoma of the prostate.
2. Age ≥ 18 years.
3. Clinically localized prostate cancer:

   * T1 (Cancer can only be seen under a microscope),
   * NX (Regional lymph nodes cannot be assessed) or N0 (Cancer cannot be seen in the lymph nodes),
   * MX (Presence of distant metastasis cannot be assessed) or M0 (Cancer hasn't spread to other parts of the body).
4. No previous treatment for prostate cancer (including hormonal therapy, radiation therapy, surgery, or chemotherapy).
5. Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1.
6. Patients must have the following laboratory values:

   1. Absolute neutrophil count (ANC) > 1500/µL
   2. Platelet count >100,000/µL
   3. Hemoglobin > 10 g/dL
   4. Bilirubin < 1.5 x upper limits of normal
   5. Aspartate aminotransferase (AST) < 1.5 x upper limits of normal
   6. Adequate estimated glomerular filtration rate (eGFR) > 30 mL/min per 1.73 m2 (adjusted for race)
7. Patient consent has been obtained according to local Institutional Review Board for acquisition of research specimens.
8. Patient is accessible and compliant for follow-up.
9. Prostate biopsy requirements:

   1. If diagnosis was within one year of baseline visit, participant must have at least one biopsy with at least 10 cores.
   2. If diagnosis was more than 1 year prior to baseline visit, participant must have a minimum of 2 biopsies, one of which must be within 2 years prior to baseline visit. Patients must have been diagnosed with prostate cancer within 2 years of randomization (no history of prostate adenocarcinoma in any biopsies taken more than 2 years prior to randomization).
10. Must have NCCN low or favorable-intermediate risk prostate cancer defined as:

    * <50% of cores involved with cancer for eligibility and 50% or greater of cores involved with cancer progression. Only cores from standard TRUS biopsy (not MRI-guided cores) will be counted towards the number of cores involved.
    * No primary Gleason pattern 4 (Gleason score 4+3) disease in any cores (TRUS or MRI-guided)
    * PSA less than 20 ng/mL
    * No extracapsular extension (<T3)
11. Patients with female partners of childbearing potential must use at least one form of Investigator-approved contraception while on-study and for 30 days after their last administration of study investigational therapy. Acceptable birth control options include:

    1. surgical sterilization (patient and/or patient's partner),
    2. approved hormonal contraceptives or therapies (such as birth control pills, Depo-Provera, or Lupron Depot),
    3. barrier methods (such as a condom or diaphragm) used with a spermicide, and
    4. an intrauterine device (IUD).

Exclusion Criteria:

1. Unwillingness or inability (such as coagulopathy) to undergo serial prostate biopsy.
2. History of other malignancies, except: adequately treated non-melanoma skin cancer or adequately treated superficial bladder cancer (Ta) or other solid tumors curatively treated with no evidence of disease for > 5 years.
3. Evidence of metastatic prostate cancer.
4. Immune-compromised patients including but not limited to: systemic immune suppressive medications within 6 weeks of enrolling; HIV-positive and below normal cluster of differentiation 4 (CD4) lymphocytes (less than 500 cells per microliter). Patients must be tested for HIV seropositivity and CD4 lymphocyte count to be eligible for the study.
5. Inability to give consent.
6. Any condition that, according to the investigator, would make the patient an inappropriate study candidate.
7. Patients with significant cardiac disease including heart failure that meets New York Heart Association (NYHA) class II and IV definitions, history of myocardial infarction within 6 months of study entry, uncontrolled dysrhythmias.
8. Patients with existing autoimmune disorders (IL-2 and GM-CSF carry risk of exacerbating underlying autoimmune disorders).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-02-28 (Estimated); Primary Completion 2021-02-28 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Prostate cancer progression measured by PSA test | At pre-study, and then every 3 months till 2 years, starting at week 7 for both arms
  Determine prostate cancer progression in patients receiving Proscavax vaccine (Arm 1) versus patients on active surveillance (Arm 2) by measuring change in PSA levels in patients in both arms
Prostate cancer progression measured by digital rectal examination (DRE) | At pre-study and then every 6-months for 2 years
  Determine prostate cancer progression in patients receiving Proscavax vaccine (Arm 1) versus patients on active surveillance (Arm 2) by performing digital rectal examination (DRE) on patients in both arms
Prostate cancer progression measured by prostate Biopsy | At pre-study and then every 12-months for 2 years
  Determine prostate cancer progression in patients receiving Proscavax vaccine (Arm 1) versus patients on active surveillance (Arm 2) by performing prostate biopsy on patients in both arms

SECONDARY OUTCOMES:
PSA doubling time | At pre-study, and then every 3 months till 2 years, starting at week 7 for both arms
  Determine the time for the PSA level to double
Assessment of Adverse Events | From first injection until 30 days past the 24-month assessments
  Confirm safety and tolerability of Proscavax vaccine

CONTACTS AND LOCATIONS:
Overall Officials: Rupal S Bhatt, MD, PhD, Principal Investigator — Harvard Medical Faculty Physicians Practice
Locations (2):
- United States (2):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts